CLINICAL TRIAL: NCT05988424
Title: Randomised Comparison of the Octaray and Pentaray Catheters
Acronym: COPEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RHM CAR0638
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Crossover from one mapping catheter to the other with randomisation as to which catheter is used first
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will not be aware which mapping catheter they are randomised to have used in their case first.
  The data will be processed for analysis blinded to the catheter used to collect the map
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentaray (Active Comparator): Initial map collected with Pentaray
  Interventions: Other: Left atrial mapping
- Octaray (Active Comparator): Initial map collected with Octaray
  Interventions: Other: Left atrial mapping

INTERVENTIONS:
Other: Left atrial mapping — Creation of a left atrial voltage map

SUMMARY:
In this study we aim to compare the mapping performance in the left atrium of the established Pentaray catheter to the newer Octaray catheter.

DETAILED DESCRIPTION:
Compared with conventional point by point mapping, the use of a multipolar high density Pentaray catheter (Biosense Webster, Diamond Bar, CA, USA) has been found to produce more rapid, accurate maps. This catheter has 20, 2mm2 electrodes. Newer, high density mapping catheters have also been introduced, capable of collecting detailed maps rapidly. Such catheters include the Orion catheter (Boston Scientific, Marlborough, MA, USA) which has 64, 0.4mm2 electrodes and has been shown to be safe and effective in real world usage, and the HD Grid (Abbott Cardiovascular, Lake Forest, IL, USA) which has 16, 1mm electrodes and has been shown to be associated with shorter procedure and fluoroscopy times and better success rates than conventional circular mapping catheters when used for AF ablation.

Of the above high density catheters, the Pentaray is integrated into the Carto3 system. An advantage of this platform for mapping is the ability to use the Tissue Proximity Indicator (TPI) Filter to reduce the number of points collected without contact and improve the accuracy of the subsequent voltage map.

A novel multipolar catheter, iterating on the previous Pentaray catheter is now being introduced: Octaray. This has 48, 0.9mm2 electrodes arranged on 8 splines. In preclinical studies, Octaray has been found to be collect maps faster, at higher density and with greater accuracy for conduction gaps than the Pentaray. The new catheter has been used safely in clinical cases.

Methods This is a randomised, prospective, single centre, interventional study, Thirty patients listed for redo AF ablation procedures on clinical grounds will be included in the study. Procedures will be under conscious sedation or general anaesthetic as per the preference of the operator, as will the mode of transeptal access and sheaths used to deliver the mapping catheter to the left atrium.

At the start of the case, two consecutive LA maps will be taken by the same operator using the Pentaray and Octaray catheters. In both cases, throughout the study the same catheter types will be used. For the Pentaray catheter, this will be the standard 4-4-4 spaced version. The Octaray for the study will be the larger, 20mm spline version, with the 3-3-3-3-3 spacing.

To minimise any learning effect from repeated map collections in the same chamber, patients will be randomly assigned, using block randomisation, as to whether their first LA map will be collected using the Octaray or Pentaray. The randomised group the patient is in will be kept in a sealed envelope which will only be opened on the day of the procedure. All maps will be respiratory gated. The same sheath will be used for both catheters. For the study protocol, maps will be taken with first one mapping catheter and then the alternative. The rhythm during collection will be the same for both maps. Ideally patients would be in sinus rhythm, with maps collected with coronary sinus pacing. If there were challenges maintaining sinus rhythm during mapping, maps can be taken in AF (though not a mixture of rhythms). The setup in terms of window of interest and references will also be identical. The map detail level will be left at 16 for all maps. The map maximum point density will be left as nominal. The fill and colour thresholds will be kept unchanged at nominal values. No ablation will be permitted between the two maps being collected. When the second map is being collected using the alternative catheter, this will be a new map and not a remap and the prior map will be hidden from the operator.

In order to control for any matrix collected by the initial catheter in taking the first map, a completely new study will be used for the second map.

TPI will be on for the entire collection period for both maps. The time when map collection was started, as well as the fluoroscopy time at that point will be noted. These values will also be noted at the end of the map collection. The aim of map collection will be to get entire coverage of the geometry with voltage data. Where this was not possible will be noted. The time for the catheter to start collecting voltage data will also be recorded, to judge the delay in TPI filter accepted points for the two catheters.

LA Map volumes will be collected from Carto3. The pulmonary veins and any left ventricle inadvertently collected will be removed from the geometries to allow quantitative assessment.

Once the mapping phase has been completed, the operator would complete the procedure as to their usual practice.

There will be no follow up needed for the study. Any acute complications will be noted - acute in this case being defined as complications occurring up to 30 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

Patients >18 years listed for redo AF ablation on clinical grounds GA or LA/sedation cases

Exclusion Criteria:

Age <18 years Pregnancy Unable or unwilling to consent Mechanical mitral valve Replacement Enrolled in another clinical study that could confound the results of this study (note: patients enrolled in complementary study are eligible for enrolment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Time to collect left atrial geometry | 1 year
  Time to collect left atrial geometry

SECONDARY OUTCOMES:
Volume of LA geometry | 1 year
  Volume of LA geometry
Map point density | 1 year
  Map point density
Time to start point collection, based on fulfilment of TPI criteria | 1 year
  Time to start point collection, based on fulfilment of TPI criteria
Low voltage area comparison | 1 year
  Low voltage area comparison
Number and size of PVI gaps identified | 1 year
  Number and size of PVI gaps identified

CONTACTS AND LOCATIONS:
Overall Officials: Waqas Ullah, Principal Investigator — University Hospital Southampton NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
Only anonymised data will be shared